CLINICAL TRIAL: NCT01676116
Title: The Efficacy of Insulin Degludec/Liraglutide in Controlling Glycaemia in Adults With Type 2 Diabetes Inadequately Controlled on GLP-1 Receptor Agonist and OAD Therapy (DUAL™ III -GLP-1 Switch)
Brief Title: The Efficacy of Insulin Degludec/Liraglutide in Controlling Glycaemia in Adults With Type 2 Diabetes Inadequately Controlled on GLP-1 Receptor Agonist and OAD Therapy
Acronym: DUAL™ III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-3851; 2012-000209-63 (EudraCT Number); U1111-1127-1321 (Other: WHO)
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; Liraglutide; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec/liraglutide + OADs (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- Liraglutide or exenatide + OADs (Active Comparator)
  Interventions: Drug: liraglutide; Drug: exenatide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Injected subcutaneously (under the skin) once daily. Dose individually adjusted. Subjects will continue their pre-trial OAD treatment without changing the frequency or dose throughout the trial.
  Arms: Insulin degludec/liraglutide + OADs
Drug: liraglutide — Subjects will continue on their pre-trial treatment of liraglutide (Victoza®) (GLP-1 receptor agonist) + OAD without changing the frequency or dose throughout the trial.
  Arms: Liraglutide or exenatide + OADs
Drug: exenatide — Subjects will continue on their pre-trial treatment of exenatide (Byetta®) (GLP-1 receptor agonist) + OAD without changing the frequency or dose throughout the trial.
  Arms: Liraglutide or exenatide + OADs

SUMMARY:
This trial is conducted in Europe, Oceania and the United States of America (USA).

The aim of the trial is to investigate the efficacy of insulin degludec/liraglutide in controlling glycaemia in adults with type 2 diabetes inadequately controlled on glucagon-like peptide-1 (GLP-1) receptor agonist and OAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus
* Glycosylated haemoglobin (HbA1c) 7.0-9.0% (53-75 mmol/mol) (both inclusive)
* Treatment with daily GLP-1 receptor agonist at maximum dose according to local label (i.e. 1.8 mg once daily (OD) Victoza® (liraglutide) or 10 microgram twice daily (BID) Byetta® (exenatide)) or documented maximum tolerated dose (i.e. 1.2 mg OD Victoza® (liraglutide) or 5 microgram BID Byetta® (exenatide)) in combination with a stable daily dose of metformin (equal to or above 1500 mg or documented maximum tolerated dose) for 90 days or more prior to screening visit (Visit 1)
* BMI (body mass index) equal to or below 40 kg/m^2

Exclusion Criteria:

* Any use of oral anti-diabetic drugs (OADs) (except for metformin, pioglitazone and sulphonylurea) for 90 days or less prior to screening visit (Visit 1)
* Use of any drug (except metformin,pioglitazone, sulphonylurea and GLP-1 receptor agonist) which in the Investigator's opinion could interfere with the blood glucose level (e.g. systemic corticosteroids)
* Treatment with any insulin regimen (short term treatment due to intercurrent illness including gestational diabetes is allowed at the discretion of the Investigator)
* Screening calcitonin equal to or above 50 ng/l
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)
* Cardiovascular disorders defined as: congestive heart failure (New York Heart Association (NYHA) class III-IV), diagnosis of unstable angina pectoris, cerebral stroke and/or myocardial infarction within the past 52 weeks prior to screening visit (Visit 1) and/or planned coronary, carotid or peripheral artery revascularisation procedures
* Proliferative retinopathy requiring acute treatment or maculopathy (macular oedema) according to the Investigator's opinion
* Subjects with a clinically significant, active (during the past 12 months) disease of the gastrointestinal, pulmonary, endocrinological (except for the type 2 diabetes mellitus), neurological, genitourinary or haematological system that in the opinion of the Investigator may confound the results of the trial or pose additional risk in administering trial products
* History of chronic pancreatitis or idiopathic acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2012-08-29 (Actual); Primary Completion 2014-03-11 (Actual); Study Completion 2014-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (98):
- United States (76):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Fair Oaks, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Tarzana, California
  - Novo Nordisk Investigational Site, Van Nuys, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Fort Myers, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Springs, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Plant City, Florida
  - Novo Nordisk Investigational Site, Winter Haven, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Arlington Heights, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Saint Charles, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Reno, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Flemington, New Jersey
  - Novo Nordisk Investigational Site, Hamilton, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, North Massapequa, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Sumter, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Jellico, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Tullahoma, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Schertz, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Orem, Utah
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Australia (5):
  - Novo Nordisk Investigational Site, Coffs Harbour, New South Wales
  - Novo Nordisk Investigational Site, Merewether, New South Wales
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, Box Hill, Victoria
  - Novo Nordisk Investigational Site, Melbourne, Victoria
- France (8):
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Boulogne-Billancourt
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Montigny-lès-Metz
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Sète
  - Novo Nordisk Investigational Site, Vénissieux
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Nyíregyhaza
  - Novo Nordisk Investigational Site, Székesfehérvár
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Lučenec
  - Novo Nordisk Investigational Site, Nitra
  - Novo Nordisk Investigational Site, Prešov

REFERENCES:
- [Result] Linjawi S, Bode BW, Chaykin LB, Courreges JP, Handelsman Y, Lehmann LM, Mishra A, Simpson RW. The Efficacy of IDegLira (Insulin Degludec/Liraglutide Combination) in Adults with Type 2 Diabetes Inadequately Controlled with a GLP-1 Receptor Agonist and Oral Therapy: DUAL III Randomized Clinical Trial. Diabetes Ther. 2017 Feb;8(1):101-114. doi: 10.1007/s13300-016-0218-3. Epub 2016 Dec 10. PMID 27943107
- [Result] Lingvay I, Handelsman Y, Linjawi S, Vilsboll T, Halladin N, Ranc K, Liebl A. EFFICACY AND SAFETY OF IDEGLIRA IN OLDER PATIENTS WITH TYPE 2 DIABETES. Endocr Pract. 2019 Feb;25(2):144-155. doi: 10.4158/EP-2018-0284. Epub 2018 Nov 1. PMID 30383495
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 81 sites in 5 countries as follows: Australia: 5 sites; France: 7 sites; Hungary: 4 sites; Slovakia 6 sites; United States: 59 sites.
Pre-assignment Details: The duration of the screening period was 2 weeks. All subjects continued GLP-1 receptor agonist and metformin±pioglitazone±SU treatments in their pre-trial doses during the screening period.
Groups:
- Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs): Subjects were treated with subcutaneous (under the skin) once daily (OD) insulin degludec/liraglutide. Treatment with insulin degludec/liraglutide was initiated at 16 dose steps containing 16 units of insulin degludec and 0.6 mg liraglutide. Adjustment of the insulin degludec/liraglutide dose was performed twice weekly based on the mean of 3 preceding daily fasting self measured plasma glucose (SMPG) values on 3 consecutive days. The aim was to achieve a fasting plasma glucose (FPG) target of 4.0-5.0 mmol/L (72-90 mg/dL) and the maximum allowed dose was 50 dose steps (50 units insulin degludec/1.8 mg liraglutide). Subjects also continued their pre-trial OADs (metformin±pioglitazone±SU) treatment without changing the frequency or dose throughout the trial, unless there was a safety concern.
- Liraglutide or Exenatide + OADs: Subjects continued on their pre-trial GLP-1 receptor agonist treatment with subcutaneous (under the skin) liraglutide (Victoza®) or exenatide (Byetta®) in stable pre-trial dose without changing the frequency or dose throughout the trial. Subjects also continued their pre-trial OADs (metformin±pioglitazone±SU) without changing the frequency or dose throughout the trial, unless there was a safety concern.
Period: Overall Study
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Started | 292 | 146
Completed | 276 | 117
Not Completed | 16 | 29
Not completed — Withdrawal criteria | 2 | 14
Not completed — Adverse Event | 1 | 2
Not completed — Unclassified | 4 | 10
Not completed — Protocol Violation | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs | Total
Number analyzed (Participants) | 292 | 146 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.9) | 58.4 (8.8) | 58.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 75 | 214
  Male | 153 | 71 | 224
HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.8 (0.6) | 7.7 (0.6) | 7.8 (0.6)
Body weight [Mean (Standard Deviation); unit: kg] | 95.6 (16.6) | 95.5 (17.3) | 95.5 (16.8)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 9 (2.1) | 9.4 (2.3) | 9.1 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline (Randomisation, Visit 2)
Time Frame: Week 0, week 26
Population: Full analysis set included all the randomised subjects. Missing values (including intermittent missing values) were imputed using the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 292 | 146
percentage of glycosylated haemoglobin | -1.32 (0.05) | -0.37 (0.07)
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) vs Liraglutide or Exenatide + OADs; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment contrast = -0.94, 95% CI 2-sided [-1.11 to -0.78]

2. Secondary Outcome: Responders Achieving Pre-defined Target: HbA1c Below 7.0% (53 mmol/Mol)
Description: Percentage of subjects achieving HbA1c below 7.0% after 26 weeks of treatment.
Time Frame: Week 26
Population: Full analysis set included all randomised subjects. Missing values (including intermittent missing values) were imputed using the last observation carried forward (LOCF) method.
Measure: Number; unit: Percentage
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 292 | 146
Percentage | 75.3 | 35.6

3. Secondary Outcome: Responders Achieving Pre-defined Target: HbA1c Below or Equal to 6.5% (48 mmol/Mol)
Description: Percentage of responders achieving pre-defined target for HbA1c - HbA1c ≤ 6.5% (48 mmol/mol).
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: Percentage
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 292 | 146
Percentage | 63 | 22.6

4. Secondary Outcome: Change From Baseline in Body Weight
Description: Mean change in body weight after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 292 | 146
kg | 2 (3.9) | -0.8 (3.0)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Mean change in fasting plasma glucose from baseline, after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: Full analysis set included all randomised subjects. A total of 430 subjects contributed to the analysis. Missing values (including intermittent missing values) were imputed using the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 285 | 145
mmol/L | -2.98 (2.28) | -0.6 (2.74)

6. Secondary Outcome: Number of Severe or Minor Hypoglycaemic Episodes
Description: Rate (events per 100 patient years of exposure) of treatment-emergent confirmed hypoglycaemic episodes. The pool of severe and minor hypoglycaemic episodes was referred to as confirmed hypoglycaemic episodes. Severe hypoglycaemia was categorised as an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as an episode with symptoms consistent with hypoglycaemia with confirmation by blood glucose <2.8 mmol/L (50 mg/dL) or PG <3.1 mmol/L (56 mg/dL), and which was handled by the subject himself/herself, or any asymptomatic blood glucose value <2.8 mmol/L (50 mg/dL) or PG value <3.1 mmol/L (56 mg/dL).
Time Frame: After 26 weeks of treatment
Population: Full analysis set included all randomised subjects. A total of 436 subjects contributed to the analysis.
Measure: Number; unit: events per 100 patient years of exposure
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 291 | 145
events per 100 patient years of exposure | 281.7 | 12.1

7. Secondary Outcome: Number of Adverse Events (AEs)
Description: Rate (events per 100 exposure years) of treatment-emergent adverse events (an event that had onset date (or an increase in severity) on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment) which occurred during the 26 weeks of treatment.
Time Frame: After 26 weeks of treatment
Population: Full analysis set included all randomised subjects. A total of 436 subjects contributed to the analysis.
Measure: Number; unit: events per 100 exposure years
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 291 | 145
events per 100 exposure years | 410.1 | 364.3

8. Secondary Outcome: Change From Baseline in Patient Reported Outcomes (PROs) Based on the Treatment Related Impact Measure - Diabetes (TRIM-D)
Description: The patient related outcome is calculated based on TRIM-D questionnaire. The TRIM-D questionnaire consists of 5 sub-domains (treatment burden, daily life, diabetes management, compliance and psychological health), where each question is scored to a 1-5-point scale with a higher score indicating a better health state (less negative impact). Mean TRIM-D individual sub-domain scores and total score are later transformed to a 0-100 scale for analysis. The mean change in scores from baseline to 26 weeks for all the individual sub domains and total scores are presented here.
Time Frame: Week 0, week 26
Population: Full analysis set included all randomised subjects. A total of 436 subjects contributed to the analysis. Missing values (including intermittent missing values) were imputed using the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 290 | 146
Scores on a scale
  TRIM-D Treatment Burden Score | 10.8 (18.8) | 5.7 (19.3)
  TRIM-D Daily Life Score | 6.3 (18.4) | 0.8 (18.2)
  TRIM-D Diabetes Management Score | 10.9 (21.3) | 4.1 (19.8)
  TRIM-D Compliance Score | 8.9 (17.3) | 4.3 (15.9)
  TRIM-D Psychological Health Score | 7.3 (14.7) | 1.4 (16.5)
  TRIM-D Total Score | 8.7 (12) | 3.1 (12.2)

9. Secondary Outcome: Change From Baseline in Patient Reported Outcomes (PROs) Based on Diabetes Treatment Satisfaction Questionnaire (DTSQ).
Description: Mean change in diabetes treatment satisfaction questionnaire (DTSQs) scores from baseline. The scores ranged from 0 to 6. Higher total score on a 0-6 point scale indicates a general higher treatment satisfaction, whereas higher score on perceived frequency of hyperglycaemia and perceived frequency of hypoglycaemia indicate that blood glucose levels are out of the target range.
Time Frame: Week 0, week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Insulin Degludec/Liraglutide + Oral Anti Diabetic Drugs (OADs) | Liraglutide or Exenatide + OADs
Number analyzed (Participants) | 290 | 146
Scores on a scale
  Treatment satisfaction scale total | 3.1 (5.6) | 1.1 (5.0)
  Hyperglycaemia | -1.8 (2.1) | -0.6 (1.9)
  Hypoglycaemia | 0.2 (1.7) | -0.1 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse events from the first trial-related activity after the subject had signed the informed consent until the end of the post-treatment follow-up period (week 27) are reported.
Description: Safety analysis set included a total of 436 subjects; (291 in the Insulin degludec/liraglutide+OADs arm and 145 in the Liraglutide or exenatide+OADs arm).
Groups:
- Insulin Degludec/Liraglutide +OADs: Subjects were treated with subcutaneous (under the skin) once daily (OD) insulin degludec/liraglutide. Insulin degludec/liraglutide was dosed on an individual basis. Subjects also continued their pre-trial OADs (metformin±pioglitazone±SU) treatment without changing the frequency or dose throughout the trial, unless there was a safety concern.
Arm/Group | Insulin Degludec/Liraglutide +OADs | Liraglutide or Exenatide + OADs
Serious Adverse Events (participants affected / at risk) | 9/291 | 3/145
Other Adverse Events (participants affected / at risk) | 88/291 | 39/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide +OADs (N=291) | Liraglutide or Exenatide + OADs (N=145)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thrombectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide +OADs (N=291) | Liraglutide or Exenatide + OADs (N=145)
Diarrhoea (Gastrointestinal disorders) | 13 (18) | 8 (9)
Headache (Nervous system disorders) | 27 (31) | 9 (14)
Lipase increased (Investigations) | 29 (31) | 7 (8)
Nasopharyngitis (Infections and infestations) | 26 (31) | 19 (20)
Upper respiratory tract infection (Infections and infestations) | 18 (18) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more public disclosures may be prepared collaboratively by the Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.